Official Study Title: The Use of New Technologies in Dentistry

NCT Number:

Document Date: May 22, 2025

## FORMULARZ ŚWIADOMEJ ZGODY

| Numer identyfikacyjny pacjenta w badaniu: |
|---|
| Ja niżej podpisany(a) oświadczam, że |
| przeczytałem/am i zrozumiałem/am powyższe informacje dotyczące opisanego badania, miałem/am |
| możliwość zadawania pytań oraz otrzymałem/am wyczerpujące, satysfakcjonujące mnie odpowiedzi |
| na zadane pytania. Wyrażam dobrowolnie zgodę na udział w tym badaniu i jestem |
| świadomy/świadoma faktu, iż w każdej chwili mogę wycofać zgodę na udział w dalszej części badania |
| klinicznego bez podania przyczyny. Przez podpisanie zgody na udział w badaniu nie zrzekam się żadnych |
| należnych mi praw. Otrzymam jedną z dwóch kopii niniejszego formularza opatrzoną podpisem i datą. |
| maicznych mi prawi o azymam jedną z dwoch kopii minejszego termalarza opaliczeną podpisem i datą. |
| Przez podpisanie tego dokumentu potwierdzam również, że zostałem/zostałam |
| poinformowany/poinformowana o sposobie przetwarzania danych z badania i że dane te będą |
| weryfikowane przez ich porównanie z moją dokumentacją medyczną oraz, że dane te są zbierane |
| jedynie w celu naukowej analizy badania. |
| Wyrażam zgodę, aby po zakończeniu tego badania moje anonimowe dane i pobrany materiał |
| biologiczny (jeśli dotyczy) były wykorzystane do kolejnych badań naukowych w celu poszerzenia wiedzy |
| w badanym obszarze: |
| □ TAK □ NIE |
| Wyrażam zgodę na przetwarzanie danych w tym badaniu zgodnie z obowiązującym w Polsce prawem |

Wyrażam zgodę na przetwarzanie danych w tym badaniu zgodnie z obowiązującym w Polsce prawem (Rozporządzenie Parlamentu Europejskiego i Rady (UE) 2016/679 z dnia 27 kwietnia 2016 r. w sprawie ochrony osób fizycznych w związku z przetwarzaniem danych osobowych i w sprawie swobodnego przepływu takich danych oraz uchylenia dyrektywy 95/46/WE). Zgadzam się na przekazanie moich anonimowych danych do innych krajów, zarówno w obrębie Europy jak i poza nią.

Dane analizowane przez władze, reprezentantów Ministerstwa Zdrowia, agencje rządowe oraz Komisje Bioetyczne dostępne będą jedynie w postaci anonimowej. Zostałem/zostałam poinformowany/poinformowana, iż w przypadku wycofania zgody na udział w badaniu zgromadzone do tej pory dane mogą zostać wykorzystane i przetwarzane jako część bazy danych badania.

Zostałem/am poinformowany/a, że zgodnie z art. 13 ogólnego rozporządzenia o ochronie danych osobowych z dnia 27 kwietnia 2016 r.:

- 1. Administratorem moich danych osobowych jest Warszawski Uniwersytet Medyczny z siedzibą w Warszawie, ul. Żwirki i Wigury 61,
- 2. Inspektorem Ochrony Danych w Warszawskim Uniwersytecie Medycznym jest Jakub Bereziewicz, nr tel. (22) 1166431, adres email jakub.bereziewicz@wum.edu.pl,
- 3. Moje dane osobowe przetwarzane będą w celu realizacji badania "Zastosowanie nowych technologii w stomatologii" w Warszawskim Uniwersytecie Medycznym na podstawie art. 9 ust. 2 lit. a ogólnego rozporządzenia o ochronie danych osobowych z dnia 27 kwietnia 2016 r.,
- 4. Moje dane osobowe mogą być ujawniane wyłącznie:
  - osobom upoważnionym u administratora do przetwarzania danych osobowych,

- podmiotom przetwarzającym na mocy umowy powierzenia,
- przedstawicielom krajowych, zagranicznych lub międzynarodowych instytucji nadzorujących badanie kliniczne po spełnieniu warunków określonych w Rozdziale V ogólnego rozporządzenia o ochronie danych osobowych z dnia 27 kwietnia 2016 r.,
- innym podmiotom upoważnionym na podstawie przepisów prawa
- 5. Moje dane osobowe przechowywane będą wyłącznie przez okres wymagany przez obowiązujące przepisy prawa,
- 6. Posiadam prawo dostępu do treści swoich danych, prawo do ich sprostowania, usunięcia, ograniczenia przetwarzania, prawo do przenoszenia danych, prawo do wniesienia sprzeciwu i prawo do cofnięcia zgody w dowolnym momencie,
- 7. Posiadam prawo wniesienia skargi do Urzędu Ochrony Danych Osobowych, gdy uzasadnione jest, że Pani/Pana dane osobowe przetwarzane są przez administratora niezgodnie z ogólnym rozporządzeniem o ochronie danych osobowych z dnia 27 kwietnia 2016 r.,
- 8. Podanie danych osobowych jest dobrowolne,
- 9. Decyzje nie będą podejmowane w sposób zautomatyzowany, nie będę podlegać profilowaniu.
- 10. Dane będą zanimizowane za pomocą nadania Pan/i numeru ID, który nie jest nigdzie przypisany do faktycznych danych osobowych.

| 11. Dostęp do danych będą mieli rea | | ektu i Wars | zawski Uniwe | rsytet Medy | czny. |
|---|---|---|---|---|---|
| Zapoznałem/zapoznałam się z warunkan wyrządzone w związku z pronumer wystawi akceptuję. | wadzeniem | badania | klinicznego | zgodnie | z poli: |
| Pacjent: | | | | | |
| lmię i nazwisko (drukowanymi literami) | Podpis | Date | a złożenia pod | pisu | |
| | (ręką pac | ienta) | | | |
| Oświadczam, że omówiłem/omówiłam zrozumiałych, możliwie prostych sformatury i znaczenia badania. | - | | | | |
| Osoba uzyskująca zgodę na badanie: | | | | | |
| Imię i nazwisko (drukowanymi literami) | Podpis | | a złożenia pod | | , |

INFORMACJA DLA PACJENTA

Tytuł badania: "Zastosowanie nowych technologii w stomatologii"

Szanowni Państwo,

Stres i lęk przed leczeniem stomatologicznym stanowi jeden z głównych problemów zdrowia

jamy ustnej w skali ogólnoświatowej. W ramach naszego projektu badamy jego poziom, aby zrozumieć

skalę problemu i jednocześnie weryfikujemy czy nowe technologie mogą ten problem rozwiązać.

Efektem tych badań będzie wniesienie nowej wiedzy do nauki oraz potencjalnie podniesienie komfortu

i satysfakcji Pana(i) z wizyty.

Jeśli zgodzi się Pan(i) wziąć udział w badaniu to oprócz standardowego zabiegu

stomatologicznego, będzie mógł(a) Pan(i) skorzystać przed i w trakcie zabiegu z nowych technologii.

Bedzie to urządzenie odtwarzające obraz i/lub dźwięk i/lub mierzące stres. Oprócz tego zbadamy

Pana(i) parametry życiowe (tetno, ciśnienie, potliwość skóry, saturację krwi) i zdiagnozujemy poziom

leku za pomocą kwestionariusza STAI (Inwentarz Stanu i Cechy Leku). Możemy również poprosić o

udzielenie informacji na temat danych społeczno-demograficznych (płeć, wiek, wykształcenie) oraz

zapytać o negatywne doświadczenia u stomatologa z przeszłości oraz czas jaki minął od ostatniej

wizyty stomatologicznej. Całość potrwa maksymalnie 10 minut. Po zakończonym zabiegu każdy

pacjent zostanie poproszony o ocenę bólu podczas wykonywanego zabiegu oraz ocenę interwencji i

jej wpływu na samopoczucie podczas wykonywanego zabiegu w grupie osób badanych. Potrwa to 5

minut. Korzyścią dla pacjentów będzie możliwość wypróbowania innowacyjnego rozwiązania jakie

daje zastosowanie nowych technologii. Natomiast ryzykiem uczestnictwa w badaniu może być

poprzez różnorodne gusta muzyczne co najwyżej uczucie irytacji.

Jednocześnie chcemy podkreślić, iż zgoda na uczestniczenie w badaniu jest całkowicie

dobrowolna i w żadnym stopniu odmowa udziału w badaniu Pana(i) nie wpłynie na opiekę

stomatologiczną. W każdym momencie trwania badania może Pan(i) zrezygnować i nie będzie to miało

wpływu na proces leczenia. Jeśli ma Pan(i) jakiekolwiek pytania dotyczące prowadzonych badań -

uprzejmie prosimy o kontakt telefoniczny z Jakubem Bereziewicz: +48 663 332 515 lub mailowy:

jakub.bereziewicz@wum.edu.pl.

## **ENGLISH TRANSLATION OF INFORMED CONSENT FORM**

| Patient identification number in the study: |
|---|
| I, the undersigned, hereby declare |
| that I have read and understood the information provided regarding the described study. I have had the opportunity to ask questions and received comprehensive and satisfactory answers. I voluntarily consent to participate in this study and I am aware that I may withdraw my consent at any time without providing any reason. By signing this consent form, I do not waive any of my legal rights. I will receive one of the two signed and dated copies of this form. |
| By signing this document, I also confirm that I have been informed about how the data from the study will be processed, that it will be verified through comparison with my medical records, and that the data is collected solely for scientific analysis of the study. |
| I agree that after the completion of this study, my anonymized data and any collected biological material (if applicable) may be used for future scientific research aimed at expanding knowledge in the studied area: |
| □ YES □ NO |
| I consent to the processing of data in this study in accordance with Polish law (Regulation (EU) 2016/679 of the European Parliament and of the Council of 27 April 2016 on the protection of natura persons with regard to the processing of personal data and on the free movement of such data). I agree to the transfer of my anonymized data to other countries, within and outside of Europe. |
| Data analyzed by authorities, representatives of the Ministry of Health, government agencies, and |

According to Article 13 of the General Data Protection Regulation of 27 April 2016:

1. The controller of my personal data is the Medical University of Warsaw, Żwirki i Wigury 61, Warsaw, Poland.

Ethics Committees will be available only in anonymous form. I have been informed that in case I withdraw my consent, data collected up to that point may still be used and processed as part of the

- 2. The Data Protection Officer at the Medical University of Warsaw is Jakub Bereziewicz, tel. +48 22 116 6431, email jakub.bereziewicz@wum.edu.pl.
- 3. My personal data will be processed for the purpose of conducting the study "Application of new technologies in dentistry" at the Medical University of Warsaw on the basis of Article 9(2)(a) of the GDPR.
- 4. My personal data may only be disclosed to:

study database.

- Persons authorized by the controller,

- Entities processing data under a data processing agreement,
- Representatives of national, foreign, or international institutions supervising the clinical trial under Chapter V of the GDPR,
- Other entities authorized under the law.
- 5. My personal data will be stored only for the period required by law.
- 6. I have the right to access my data, rectify, delete, restrict processing, transfer, object, and withdraw consent at any time.
- 7. I have the right to lodge a complaint with the Data Protection Authority if I believe my data is being processed unlawfully.
- 8. Providing personal data is voluntary.
- 9. Decisions will not be made automatically and I will not be subject to profiling.
- 10. Data will be anonymized using an ID number not linked to personal data.
- 11. Access to data will be granted to project implementers and the Medical University of Warsaw.

| I have reviewed and accepted the damages resulting from the clinic | | , |
|---|---|---|
| number | issued by | Insurance Company. |
| Patient: | | |
| Full name (printed) | Signature | Date |
| (pa | tient's own hand) | |
| I declare that I have discussed the study with the patient using understandable, simple language and provided information on the nature and significance of the study. | | |
| Person obtaining consent: | | |
| Full name (printed) | Signature | Date |

## **ENGLISH TRANSLATION OF PATIENT INFORMATION SHEET**

Title of the study: "Application of new technologies in dentistry"

Dear Participant,

Stress and anxiety related to dental treatment are among the most significant global oral health issues. In this project, we examine the level of such stress to understand the scale of the problem and evaluate whether new technologies can help address it. The study aims to contribute new scientific knowledge and potentially enhance your comfort and satisfaction with dental visits.

If you agree to participate, you will undergo a standard dental procedure while also having the opportunity to use innovative technologies before and during the treatment. This may include a device that displays images and/or sound and/or measures stress. We will also monitor your vital signs (heart rate, blood pressure, skin conductance, blood oxygen saturation) and assess anxiety levels using the STAI (State-Trait Anxiety Inventory). We may also ask for socio-demographic data (gender, age, education), past negative dental experiences, and the time since your last dental visit. This part will take a maximum of 10 minutes. After the procedure, you will be asked to rate pain experienced and the impact of the intervention on your well-being, taking about 5 minutes. Benefits include trying innovative technologies; the only potential risk is mild irritation due to personal preferences.

Participation is entirely voluntary. Refusal will not affect your dental care. You may withdraw at any point without consequences. For any questions, contact Jakub Bereziewicz at +48 663 332 515 or jakub.bereziewicz@wum.edu.pl.

Project implementers: Dr. hab. n. med. Jan Kowalski and Jakub Bereziewicz